CLINICAL TRIAL: NCT06441721
Title: Vitamin b12 Deficency and Its Impact on Chronic Haemodialysis Patient and Its Effect on Anemia and Neuropathy
Brief Title: Vitamin B12 Status and Its Impact on Chronic Haemodialysis Patient
Acronym: Haemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Afaf Bakry Amin Omer, Doctor, Assiut University
Other Study IDs: Vitamin B12 and Haemodialysis
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease on Dialysis; Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vitamin b12 measure — Measure vitamin b12 in serum and its impact on Haemodialysis patient

SUMMARY:
To evaluate vitamin B12 level in haemodialysis patients and its impact on hematological and neurological manifestations

DETAILED DESCRIPTION:
Vitamin B12 (cobalamin) is a water-soluble vitamin involved in several normal cellular functions (1). Vitamin B12 is required for the development, myelination, and function of the central nervous system; healthy red blood cell formation; and DNA synthesis (2- 4). Low levels of vitamin B12 have been associated with high concentrations of homocysteine (Hcy) and can lead to health complications (5). Hyperhomocysteinemia is an important risk factor for cardiovascular disease (6). Vitamin B12 and other B vitamins are involved in homocysteine metabolism, and researchers have hypothesized that supplementation with these micronutrients can reduce the risk of cardiovascular disease by lowering homocysteine levels (7, 8). Vitamin B12 deficiency is one of the causes of Macrocytic anaemia with increased mean corpuscular volume (MCV), defined as more than 100 fL, which is the hallmark of megaloblastic anaemia

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease on haemodialysis pts.
* Parients more than 18 years .
* CKD patients controled group stage 3and stage 4.

Exclusion Criteria:

* Recent renal transplantation patients.
* Patients on sulpha drugs.
* Patients on methotrexate.
* Patients on anticonvulsant.
* Patients on chemotherap agent.
* Patients on colchicine.
* Patients on bile acid sequestrant.
* Patients on h2blockers.
* Patients on metformin.
* Patients on proton pump inhibitors .
* Diabetic patients.
* Parients with history of intestinal surgery.
* Patients diagnosed with malabsorption syndrome.
* Patient on vitamin b12 intake.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: evaluate vitamin b12 in serum in chronic haemodialysis patient not diabetic age group 18-80 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
vitamin b12 in serum | one year
  vitamin b12 evaluation vitamin b12 evaluation

REFERENCES:
- [Background] Juszczak AB, Kupczak M, Konecki T. Does Vitamin Supplementation Play a Role in Chronic Kidney Disease? Nutrients. 2023 Jun 23;15(13):2847. doi: 10.3390/nu15132847. PMID 37447174
- [Result] Fahndrich C, Gemperli A, Baumberger M, Harder M, Roth B, Schaefer DJ, Wettstein R, Scheel-Sailer A. Risk factors of major complications after flap surgery in the treatment of stage III and IV pressure injury in people with spinal cord injury/disorder: a retrospective cohort study. Spinal Cord. 2024 Jan;62(1):34-41. doi: 10.1038/s41393-023-00944-9. Epub 2023 Dec 20. PMID 38123748
- See also: Annual dialysis data report 2015 jsdt renal data — http://doi.org/10.1186/s41100-018-0149-8